CLINICAL TRIAL: NCT02434133
Title: Cross Sectional Study of Vaccine Antibody Response in Inflammatory Bowel Disease Patients
Status: Completed | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Other Study IDs: 2015-0340; Tetanus/MMR (Other: UW-Madison Study Staff)
Record Dates: First submitted 2015-04-27; First posted 2015-05-05 (Estimated); Last update posted 2018-11-27 (Actual); Status verified 2018-11

CONDITIONS: Inflammatory Bowel Disease (IBD)
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood sample to measure antibody concentration
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Case (Group A): Group A (Immunomodulator) currently taking azathioprine or 6- mercaptopurine (Blood Draw)
  Interventions: Procedure: Blood Draw/Data Collection
- Case (Group B): Group B (Biologic group) currently taking anti-TNF therapy (infliximab, golimumab, adalimumab, or certolizumab).
  (Blood Draw)
  Interventions: Procedure: Blood Draw/Data Collection
- Case (Group C): Group C (Combination therapy) currently taking anti-TNF therapy and an immunomodulator (including methotrexate) (Blood Draw)
  Interventions: Procedure: Blood Draw/Data Collection
- Control: Individuals will be obtained from patients without an IBD diagnosis coming to Digestive Health Center for endoscopic procedures or clinic visits.
  (Blood Draw)
  Interventions: Procedure: Blood Draw/Data Collection

INTERVENTIONS:
Procedure: Blood Draw/Data Collection — Participation will involve an extra 8ml tube of blood and a review of their medical records for medications and immunization history.

SUMMARY:
The investigators proposed study is the first of its kind. The investigators will measure measles, mumps, rubella, tetanus, diphtheria and pertussis antibodies in patients on the current IBD treatment modalities and compare the vaccine antibody concentrations and correlate them with time since immunization.

DETAILED DESCRIPTION:
Tetanus and diphtheria have become rare diseases because of widespread immunization that began during World War II. The percentage of people who got pertussis (whooping cough) also went down after vaccination, but large outbreaks have occurred over the past decade. Measles, mumps, rubella (German measles) and varicella (chicken pox) are illnesses that resolve quickly, but which can cause other diseases to take hold or get worse. Routine vaccination can prevent infection and has been and recommended for use in the United States beginning in the 1960s and 1970s; and in 1995 for varicella. Today measles, mumps, and rubella are especially uncommon in the U.S. thanks to vaccination programs; and the percentage of people with varicella is going down. Despite widespread vaccination efforts, there have been recent outbreaks of measles and mumps in the U.S., in part because these diseases are still common in other parts of the world.

Inflammatory bowel disease (IBD) is a chronic inflammatory disorder of the gastrointestinal tract which includes Crohn's disease (CD) and ulcerative colitis (UC). Treatment options for IBD consist of immunosuppressive therapy, meaning that the drugs weaken the immune system, such as systemic corticosteroids, immunomodulators (thiopurines and methotrexate) and/or biologics, such as tumor necrosis factor alpha (TNF) agents or an integrin inhibitor (vedolizumab). Patients with IBD can achieve clinical remission and decrease the risk of complications with treatment; however, treatment can also increase the risk for infections because they weaken the immune system. Some of these infections are preventable with routine vaccination.

You are invited to take part in this research project to determine if people with IBD on different types of therapy have a lower amount of antibodies than healthy individuals. Antibodies are proteins used by the immune system to attack viruses like tetanus and measles. Antibodies can be introduced into the body through vaccines. The fewer antibodies there are, the harder it is for the antibodies to attack a virus, meaning that the person could get sick with a virus. This research project will help us figure out whether people with IBD have fewer antibodies than people without IBD. The investigators will also look at whether the type of treatment people take for IBD affects the amount of antibodies. T

This will tell us who is more likely to get sick from viruses, and why. The investigators will recruit 90 IBD patients under treatment for their IBD as well as 20 healthy controls for a total of 110 patients at the University of Wisconsin Hospital & Clinics.

ELIGIBILITY:
Inclusion Criteria

* A history of chronic (greater than 3 month) ulcerative colitis or Crohn's disease diagnosed and documented by the standard clinical, radiographic, endoscopic and histopathologic criteria.
* Undergoing blood work the day of the study visit for routine blood monitoring due to medication.
* Has a documented tetanus-diphtheria (Td) or tetanus-diphtheria-acellular pertussis (Tdap) in the Wisconsin Immunization Registry (WIR) at least 4 weeks prior to entering study.
* Has a document measles, mumps and rubella (MMR) in the Wisconsin Immunization Registry (WIR) at least 4 weeks prior to entering study. This will need to be met by 50% of patient in group A-C.
* Is currently taking one of the following medication regimens for at least 3 months.
* Group A (Immunomodulator) currently taking azathioprine or 6- mercaptopurine
* Group B (Biologic group) currently taking anti-TNF therapy (infliximab, golimumab, adalimumab, or certolizumab).
* Group C (Combination therapy) currently taking anti-TNF therapy and an immunomodulator (including methotrexate)
* The patient must understand and voluntarily sign the informed consent document.

Exclusion Criteria

* Unconfirmed Td or Tdap vaccination status
* Patients in whom venipuncture are not feasible due to poor tolerability or lack of easy access.

CONTROLS Inclusion Criteria

* Has a documented tetanus-diphtheria (Td) or tetanus-diphtheria-acellular pertussis (Tdap) in the Wisconsin Immunization Registry (WIR) at least 4 weeks prior to entering study.
* Has a document measles, mumps and rubella (MMR) at least two injections in the Wisconsin Immunization Registry (WIR) at least 4 weeks prior to entering study.

CONTROLS Exclusion Criteria

* Currently on immunosuppressive therapy
* Has a chronic health condition that may have an impact on vaccine antibody concentrations as deemed by the investigators, including chronic liver disease, celiac disease, history of solid organ or bone marrow transplantation.
* Older than age 65 years
* Unconfirmed MMR vaccination status
* Patients in whom venipuncture are not feasible due to poor tolerability or lack of easy access.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The subject population will consist of individuals with inflammatory bowel disease and healthy controls.
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2015-04; Primary Completion 2016-04 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
To compare antibody concentrations and seroprotection rates | 12 month study
  To compare tetanus, diphtheria, and pertussis antibody concentrations and seroprotection rates in patients with IBD treated with combination therapy to healthy individuals.
To compare antibody concentrations and seroprotection rates | 12 month study
  To compare measles, mumps, and rubella antibody concentrations and seroprotection rates in patients with IBD treated with combination therapy to healthy individuals.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Wisconsin Hospital & Clinics, Madison, Wisconsin, United States

REFERENCES:
- [Derived] Caldera F, Misch EA, Saha S, Wald A, Zhang Y, Hubers J, Megna B, Ley D, Reichelderfer M, Hayney MS. Immunosuppression Does Not Affect Antibody Concentrations to Measles, Mumps, and Rubella in Patients with Inflammatory Bowel Disease. Dig Dis Sci. 2019 Jan;64(1):189-195. doi: 10.1007/s10620-018-5321-z. Epub 2018 Oct 13. PMID 30317494
- [Derived] Caldera F, Saha S, Wald A, Garmoe CA, McCrone S, Megna B, Ley D, Reichelderfer M, Hayney MS. Lower Sustained Diphtheria and Pertussis Antibody Concentrations in Inflammatory Bowel Disease Patients. Dig Dis Sci. 2018 Jun;63(6):1532-1540. doi: 10.1007/s10620-018-5043-2. Epub 2018 Mar 29. PMID 29594970